CLINICAL TRIAL: NCT05286489
Title: Effects of Selected Exercise Program on Microcirculation and Lymphedema in Postmastectomy Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Mohamed othman, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00000001
Record Dates: First submitted 2022-03-01; First posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Mastectomy; Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): Qigong exercise program twice weekly for 8 weeks postmastectomy in addition to traditional medical and physical therapy treatment.
  Interventions: Combination Product: Qigong exercise
- group B (Other): traditional medical and physical therapy treatment only .
  Interventions: Combination Product: Qigong exercise

INTERVENTIONS:
Combination Product: Qigong exercise — The qigong style they learned is known as 18 Forms Tai Chi Internal Qigong. It is a kind of physical and mental exercise (internal qigong) that focuses on relaxation, deep breathing, and slow and coordinated movements and uses the mind to guide these movements. There are a total of 18 upper and lower body movements, and all of the techniques are performed while either standing or semi squatting. qigong practice session was initiated immediately and continued for about 6 minutes. Each participant in the qigong group performed 18 Forms Tai Chi Internal Qigong once and was assessed immediately afterward in sitting (to measure the vascular outcomes) and lying (to measure the upper limb circumference) positions. The control participants were given no specific exercise instruction after the baseline assessment. Instead, they were asked to rest (sit quietly in the laboratory) for 6 minutes and then participated in the postassessment directly

SUMMARY:
PURPOSE: to assess the efficacy of Qigong exercise on microcirculation in postmastectomy lymphedema patient.

BACKGROUND: Qigong is a mind-body integrative exercise originating from traditional Chinese medicine and is used to improve health and energy levels through regular training, yet its effects are not empirically assessed.

Qigong may be a potentially beneficial exercise for survivors of breast cancer and could be used to regulate upper limb blood flow and decrease lymphedema. There is lack in knowledge and information in published studies about the efficacy of Qigong exercise on microcirculation in postmastectomy lymphedema patient.

So, this study will be designed to provide a guideline about the efficacy of Qigong exercise on microcirculation in postmastectomy lymphedema patient.

HYPOTHESES:

It will be hypothesized that:

It was hypothesized that Qigong exercise has no or limited effect in microcirculation in postmastectomy lymphedema patient.

RESEARCH QUESTION: Does Qigong exercise an effect on microcirculation in postmastectomy lymphedema patient?

DETAILED DESCRIPTION:
1. Measurement procedure:

   Both methods of measurements will be done before the beginning of the treatment (pre-treatment) then at the end of the study after 2 months of treatment (post treatment) for both groups of the study.

   A-Upper Limb Circumference by manual goniometer

   B- LASER Doppler Imaging:
2. Treatment procedures:

In this study the treatment protocol was presented in the form of an exercise program lasted for 60 minutes, twice weekly for 8 weeks postmastectomy and achieved under the following phases:

1. Warming up phase:

   The main aim of this phase was to get the muscles warm and loose for strength training. The subject has to train for ten minutes aerobic exercise at a mild velocity before the beginning of each exercise session. Warming up helps direct needed blood flow to the muscles and prepares the body for exercise. Warming up is important for preventing injury as well as gaining maximal benefit from the exercise, because loose and warm muscles respond better to the challenge of the program.
2. Exercise phase:

Participants in the experimental group were qigong practitioners. The qigong style they learned is known as 18 Forms Tai Chi Internal Qigong, which is quite popular among Chinese breast cancer patients. It is a kind of physical and mental exercise (internal qigong) that focuses on relaxation, deep breathing, and slow and coordinated movements and uses the mind to guide these movements. There are a total of 18 upper and lower body movements, and all of the techniques are performed while either standing or semi squatting. Qigong practice session was initiated immediately and continued for about 6 minutes. Each participant in the qigong group performed 18 Forms Tai Chi Internal Qigong once and was assessed immediately afterward in sitting (to measure the vascular outcomes) and lying (to measure the upper limb circumference) positions. The control participants were given no specific exercise instruction after the baseline assessment. Instead, they were asked to rest (sit quietly in the laboratory) for 6 minutes and then participated in the post assessment directly

ELIGIBILITY:
Inclusion Criteria:

* age from 25-40 years
* with or without adjuvant chemotherapy/ radiotherapy
* had completed conventional treatments of breast cancer
* medically stable
* had lymphedema, defined as a circumference difference greater than 2 cm at any point between the surgical-side upper limb and the contralateral upper limb
* had no known neurological deficit resulting from breast cancer treatment.
* Participants were also able to perform 18 Forms Tai Chi Internal Qigong independently.

Exclusion Criteria: Participants were excluded if they:

* had significant neurological, musculoskeletal, cardiovascular, peripheral vascular, or kidney disorders.
* had recurrent breast cancer or cancer in another organ during the study period.
* did regular exercises other than qigong
* smokers
* received lumpectomy but not mastectomy
* pregnant during the study period.

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — as the study for post mastectomy patients it's relevant for 1%
Enrollment: 30 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
microcirculation of blood cells | changes from the baseline at 2 months after treatment
  * As these blood cells are moving, the reflected light is subject to the Doppler shift, which is a small change in frequency.
  * When laser light penetrates the tissue under study it is scattered and partly absorbed. Some of the scattered light returns to the tissue surface, where it is registered by a photo detector inside the instrument. This signal is then processed to extract information about the microcirculatory blood flow. According to the Doppler principle, light particles which hit moving blood cells undergo a change in wavelength/frequency (a Doppler shift), while light particles which encounter static structures return unchanged. The perfusion can be calculated since the magnitude and frequency distribution of the doppler shifted light are directly related to the number and velocity of blood cells but unrelated to their direction of movement.
Upper Limb Circumference | changes from the baseline at 2 months after treatment
  The circumferences of both arms that represented the participants' lymphedema status were taken at the level of (a) 10 cm proximal to the lateral epicondyle; (b) the elbow joint, right at the lateral epicondyle; (c) 10 cm distal to the lateral epicondyle; and (d) the wrist joint, just distal to the ulnar styloid process. The upper limb circumferences were measured with a cloth measuring tape. The difference in each circumference measurement between the ipsilateral and contralateral arms was calculated to detect a 2 cm between-side difference.

CONTACTS AND LOCATIONS:
Overall Officials: eman othman, PhD, Study Chair — assistant professor at faculty of physical therapy, Cairo university
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in bee venom or ulcer . we will share the results of this study within 1 year following publication.
Supporting Information: SAP, ICF
Time Frame: 1 year after publication
Access Criteria: the criteria will be assessed by the publication of the trial in an international journals.